CLINICAL TRIAL: NCT07058103
Title: Efficacy and Safety of Tislelizumab in Combination With Cyclophosphamide, Mitoxantrone Liposomes, Chidamide, and Prednisone in the Treatment of R/R AITL: a Multicenter, Single-arm, Prospective Clinical Study
Brief Title: Tislelizumab , Cyclophosphamide, Mitoxantrone Liposomes, Chidamide, and Prednisone in the Treatment of R/R AITL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2025-KL113-02
Record Dates: First submitted 2025-06-10; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Angioimmunoblastic T-Cell Lymphoma Recurrent; Angioimmunoblastic T-Cell Lymphoma Refractory
MeSH Terms: interventions — tislelizumab; Cyclophosphamide; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with relapsed/refractory angioblastic T cell lymphoma (Experimental): Patients with relapsed/refractory angioblastic T cell lymphoma
  Interventions: Drug: tislelizumab in combination with cyclophosphamide, mitoxantrone liposomes, chidamide, and prednisone

INTERVENTIONS:
Drug: tislelizumab in combination with cyclophosphamide, mitoxantrone liposomes, chidamide, and prednisone — tislelizumab: 200mg on d1 every 3 weeks; chidamide: 20mg twice a week at least 3 days apart; cyclophosphamide: 750mg/m2 on Day 1 of each cycle, every 4 weeks; mitoxantrone liposomes: 20mg/m2 on Day 1, every 4 weeks; prednisone: 100mg/day on Day 1 to Day 5 of each course, every 4 weeks.

SUMMARY:
Angioimmunoblastic T cell lymphoma (AITL) is a rare and aggressive lymphoma. Some patients relapsed after initial treatment or did not respond to standard treatment (refractory). Subsequent treatment options are limited and the efficacy is not ideal. This study attempts to explore the possibility of improving the efficacy of immunotherapy combined with chemotherapy and epigenetic regulatory drugs.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of AITL according to WHO classification in 2016, and pathological diagnosis of AITL according to WHO classification in 2016, and at least one evaluable or measurable lesion meeting Lugano2014 criteria: lymph node lesion, detectable lymph node length>1.5cm; non-lymph node lesion, detectable extra-nodal lesion length>1.0cm;
* Refractory or relapsed after at least one systemic therapy (including chemotherapy, stem cell transplantation)*;
* Age ≥18 years old, male or female, ECOGPS≤3 points;
* Life expectancy exceeds 3 months;
* Follow-up conditions. Patients understand the characteristics of the disease and voluntarily join the study protocol for treatment and follow-up.

  * : Relapse: patients achieve complete response (CR) or partial response (PR), disease progression (PD) ≥6 months; refractory: treatment failure (no PR) or PD <6 months after the last chemotherapy.

Exclusion Criteria:

Subjects who meet any of the following criteria are not eligible for inclusion in this study:

* Patients with abnormal liver and kidney function, specifically serum direct bilirubin, serum indirect bilirubin and/or alanine aminotransferase, aspartate aminotransferase and serum creatinine>2 times normal values, unless abnormal liver and kidney function is considered to be related to lymphoma;
* Bone marrow failure, specifically defined as absolute neutrophil count (ANC)<1.5*10^9/L or platelets <75*10^9/L or Hb<90g/L, unless changes in hemogram are considered to be associated with lymphoma infiltration of the bone marrow;
* The subject's prior history of antineoplastic therapy meets one of the following conditions: (1) prior mitoxantrone or mitoxantrone liposome therapy;(2) prior PD-1 or PD-L1 inhibitor therapy;(3) Angioimmunoblastic T-cell lymphoma previously treated with histone deacetylase inhibitors;
* Chronic heart failure with cardiac function class III or IV; or left ventricular ejection fraction <50%; or patients with the following cardiac diseases within 6 months: acute coronary syndrome; acute heart failure (Class III or IV of cardiac function class); patients with a history of clinically significant QT prolongation (>450 ms for men,>470 ms for women), ventricular tachycardia (VT), atrial fibrillation (AF), heart block, symptomatic coronary heart disease requiring medical treatment;
* AIDS, syphilis, active B (HBV DNA>1*10^4 copies/ml) and hepatitis C;
* Patients with other malignancies that are not effectively controlled; or with other hematological disorders (e.g. hemophilia, myelofibrosis, etc.), the investigator considers that the patient is not suitable for enrollment;
* History of autoimmune disease, receiving immunosuppressive therapy before enrollment, immunosuppressive dose>10 mg/day or oral prednisone for more than 2 weeks;
* Clinically uncontrolled active infection (including bacterial, fungal or viral infections), and drug therapy is ineffective;
* Patients with uncontrolled hemophagocytic syndrome;
* Patients who have received secondary surgery or above within 3 weeks before treatment;
* Patients who have participated in clinical trials of other drugs within 30 days before enrollment or are participating in clinical trials of other new drugs;
* Pregnant and lactating women and patients of childbearing age who are unwilling to take contraceptive measures;
* Known allergies to investigational drug components;
* The investigator considers that the enrollment is not suitable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the Objective Response Rate (Complete response+Partial response) of tirelizumab in combination with cyclophosphamide, mitoxantrone liposomes, sidaraniline, and prednisone in subjects with relapsed/refractory angioimmunoblastic T-cell lymphoma | Time forecasting: 24 months

SECONDARY OUTCOMES:
24-month Overall Survival Rate in relapsed/refractory AITL | From first dose until death from any cause (assessed at 24 months)
  Proportion of patients alive at 24 months after initiation of tirelizumab combination therapy
24-month Progression-free Survival Rate in relapsed/refractory AITL | From first dose until first documented progression or death (assessed at 24 months)
  Proportion of patients without disease progression at 24 months per Lugano 2014 criteria
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Time forecasting: 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China